CLINICAL TRIAL: NCT00859495
Title: Phase II, A Study of Lung-Sparing Combined Modality Protocol for the Treatment for Malignant Pleural Mesothelioma: The Columbia Protocol
Brief Title: Trimodal Lung-Sparing Treatment of Pleural Mesothelioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAB9658
Record Dates: First submitted 2009-03-09; First posted 2009-03-11 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Doxorubicin; liposomal doxorubicin; Cisplatin; Pemetrexed; Radiotherapy; ING2 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Multimodal lung sparing regimen (Experimental): Intrapleural chemotherapy plus systemic chemotherapy:
  Thoracoscopy to implant two intrapleural catheters followed by intrapleural chemotherapy with doxorubicin and cisplatin (weeks 1, 2, 4, 5, 7, and 8). Systemic chemotherapy treatments with cisplatin and pemetrexed during weeks 3, 6, and 9. Intrapleural radiotherapy with P-32 will be given 3 weeks after last dose of chemotherapy and 11 to 12 weeks after initial thoracoscopy.
  Interventions: Drug: Doxorubicin; Drug: Cisplatin; Drug: Pemetrexed; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Doxorubicin — A medication used in cancer chemotherapy, derived by chemical semisynthesis from a bacterial species.
  Other Names: Doxil
Drug: Cisplatin — Platinum-based antineoplastic
  Other Names: Cisplatinum; Platinol
Drug: Pemetrexed — Folate Analog Metabolic Inhibitor
  Other Names: Alimta
Radiation: Radiotherapy — Standard procedure given 3 weeks after last dose of chemotherapy
  Other Names: Intrapleural radiotherapy with P-32

SUMMARY:
The primary objective of the study is to determine the feasibility (as determined by lack of serious adverse events) and tolerability (as determined by patient's ability to complete the study) of a multimodal lung sparing regimen of surgery, interpleural and intravenous chemotherapy, and local P-32 irradiation for malignant pleural mesothelioma.

DETAILED DESCRIPTION:
Current surgical and/or chemotherapeutic approaches for malignant pleural mesothelioma are unsatisfactory and have not been shown to significantly prolong survival, and often lead to worsened pulmonary function and quality of life. We will investigate whether a prospective trial of trimodal (surgery, pleural chemotherapy, and pleural radiation) therapy can improve the overall 1 year survival in patients with malignant pleural mesothelioma. The proposed treatment will include exploratory thoracoscopy, placement of Mediport catheters into the pleural space, intraoperative chemotherapy, repeated intraperitoneal chemotherapy, and intrapleural instillation of radioactive P32 to radiate the pleural surfaces. In addition, because this study is randomized, half the patients will receive an additional three intravenous systemic chemotherapy treatments of cisplatin and pemetrexed (Alimta) in tandem with their intrapleural chemotherapy (weeks 3, 6, and 9 only).

The potential significance of this research is that such treatment may render it less necessary to surgically remove the affected lungs in whole or in part, in order to achieve significant disease cytoreduction. We hope to alter the currently accepted paradigm that major lung surgery is an inescapable component of such treatment, and advance the concept that a combination of judicious preparative surgery, systemic chemotherapy, and locoregional drug treatment of the pleural surfaces may offer the best hope for prolongation of survival with intact lung function.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant mesothelioma, < 20% sarcomatoid type
* No radiographic or other imaging evidence of Stage IV (cardiac, mediastinal, peritoneal, other distant) disease.
* Ineligible for other high priority national or institutional study.
* Age >18 years [to physiologic 75 years].
* Life expectancy > 3 months.
* Performance status, PS 0-2 [Karnofsky Performance Status, KPS=70-100 %].
* Prior therapy allowed (one prior systemic regimen) meeting the following parameters.
* No prior chest radiation therapy within 6 weeks of treatment
* No prior chemotherapy regimens within four weeks of treatment
* Non pregnant, non-lactating. (serum HCG test will be performed in patients in whom there is a possibility of pregnancy.)
* Required initial laboratory data/clinical parameters (see also Sec. 8.0) White cell count: >3000/ul. Platelet count: >100,000/ul. Creatinine clearance: ≥ 45 ml/min Bilirubin: < 2 x ULN SGOT or SGPT: < 2 x ULN
* Informed Consent: Each patient must be completely aware of the nature of his/her disease process and must willingly give consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts.
* No other coexistent malignancy. However, curatively treated or fully controlled solid tumors (other than mesothelioma) may be eligible if in the judgement of the PI, the benefit of treatment outweighs the risk.
* No serious medical or psychiatric illness preventing informed consent or intensive treatment (e.g., serious infection, congestive heart failure, angina pectoris, cardiac arrhythmia(s), or uncontrolled hypertension). HIV status or other severe illnesses will be assessed using medical records.

Exclusion Criteria:

* If any of the inclusion criteria was not met.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert N Taub, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Multimodal Lung Sparing Regimen: Intrapleural chemotherapy plus systemic chemotherapy:
  Thoracoscopy to implant two intrapleural catheters followed by intrapleural chemotherapy with doxorubicin and cisplatin (weeks 1, 2, 4, 5, 7, and 8). Systemic chemotherapy treatments with cisplatin and pemetrexed during weeks 3, 6, and 9. Intrapleural radiotherapy with P-32 will be given 3 weeks after last dose of chemotherapy and 11 to 12 weeks after initial thoracoscopy.
  Doxorubicin: A medication used in cancer chemotherapy, derived by chemical semisynthesis from a bacterial species.
  Cisplatin: Platinum-based antineoplastic
  Pemetrexed: Folate Analog Metabolic Inhibitor
  Radiotherapy: Standard procedure given 3 weeks after last dose of chemotherapy
Period: Overall Study
Arm/Group | Multimodal Lung Sparing Regimen
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Multimodal Lung Sparing Regimen
Number analyzed (Participants) | 9
Age, Customized [Count of Participants; unit: Participants]
  18-65 years | 7
  > 65 years | 2
Sex/Gender, Customized [Count of Participants; unit: Participants] — Data were not collected.
  Participants
    Non-specific | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 8
  Hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Were Able to Complete Trimodal Therapy (Combination of Surgery, Intrapleural and Systemic Chemotherapy and P-32 Radiotherapy).
Description: To determine the feasibility of multimodal lung sparing regimen. Intrapleural chemotherapy (12 weeks) will be administered within two weeks after surgery. Approximately 30 days post last dose of chemotherapy (+/- 14 days), the patient should be reassessed for resolution of any treatment-related toxicity which may have occurred during the course of study participation.
Time Frame: 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Multimodal Lung Sparing Regimen
Number analyzed (Participants) | 9
Participants | 9

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Multimodal Lung Sparing Regimen
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
Study was terminated early due to the retirement of the study physician responsible for the P-32 radiotherapy, and the need for further funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes